CLINICAL TRIAL: NCT04687098
Title: Risk-adapted Therapy for Primary Acute Myeloid Leukemia (AML) in Adult Patients up to 70 Years Old
Brief Title: Risk-adapted Therapy for Primary Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Cooperativo de Estudio y Tratamiento de las Leucemias Agudas y Mielodisplasias (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AML-12
Record Dates: First submitted 2020-12-18; First posted 2020-12-29 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Leukemia; Myeloid
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — Idarubicin; Cytarabine; Granulocyte Colony-Stimulating Factor; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Risk-adapted postremission treatment. (Other): Induction (idarubicin, cytarabine), first consolidation (high dose cytarabine), risk- stratification: allogeneic matched related or unrelated donor transplant vs. consolidation courses.
  Interventions: Drug: Idarubicin; Drug: Ara-C; Drug: G-CSF; Procedure: Allogeneic matched or unrelated donor transplant.; Procedure: Autologous peripheral blood stem cell transplant; Procedure: Measurable residual disease

INTERVENTIONS:
Drug: Idarubicin — 12 mg/m2/day; intravenous, administration at induction phase, days 1 to 3.
  Other Names: Ida
Drug: Ara-C — 200mg/m2/day, intravenous at induction phase; days 1-7.
  - High dose during consolidation phase. In patients up to 60 years 3g/m2/12hours days 1,3,5, and patients 60 to 70 years: 1.5g/m2/12hours days 1,3,5.
  Other Names: HDAC
Drug: G-CSF — * Administration at induction phase to remission days 1 to 7. G-CSF will not be initiated if the leukocyte count is over 30x10e9/L at diagnosis or will be interrupted if the leukocyte count during treatment arises 30x10e9/L.
  * Administration at consolidation phase day 7.
  Other Names: Pegfilgrastim
Procedure: Allogeneic matched or unrelated donor transplant. — To be performed in patients in the intermediate or adverse risk groups.
Procedure: Autologous peripheral blood stem cell transplant — To be considered in patients in the intermediate risk group without an available allogeneic donor and negative measurable residual disease, per center decision.
Procedure: Measurable residual disease — To be performed either with molecular monitoring or, if not applicable, by flow cytometry. Pre-stablished cut-off values are defined for decision-making.
  Other Names: MRD

SUMMARY:
The AML-12 study investigates the efficacy and toxicity of standard induction chemotherapy with idarubicin and cytarabine (IC) with G-CSF priming followed by a risk-adapted post remission therapy for patients up to the age of 70 diagnosed with de novo acute myeloid leukemia (AML).

Modifications from the previous protocol AML-03 (NCT01723657) include removal of etoposide in induction, limitation of the GCSF priming to the induction phase and categorization of post remission therapy (stem cell transplant or 2 high dose cytarabine consolidations) according to diagnostic genetics as well as post-remission clearance of measurable residual disease.

The aims of these modifications are to improve the overall survival and leukemia free survival of acute myeloid leukemia patients with a risk-adapted approach.

DETAILED DESCRIPTION:
Induction chemotherapy: Idarubicin (12mg/m2/day intravenous, days 1-3), Low-dose cytarabine (200mg/m2/day, intravenous in continuous infusion, days 1-7) and G-CSF priming 150mcg/m2/day, subcutaneous from day 0 to the last day of chemotherapy if white blood cell count (WBC) <30x10E9/L.

This induction chemotherapy can be repeated twice in the case of partial response (PR) to achieve complete response (CR).

Once CR is achieved (with one or two induction cycles), all patients receive a consolidation course with high-dose cytarabine (3000mg/m2/12h days 1, 3 and 5) and pegfilgrastim 6mg on day 6.

After this, patients will be allocated to the different risk groups as follows:

* Favorable risk group [patients with t(8;21)(q22;q22)/RUNX1/RUNX1T1, inv(16)(p12;q22) or t(16;16)/CBFB/MYH11; Intermediate risk cytogenetics (MRC 2010) and NPM1 mutation with FLT3 wild type or low ratio of FLT3 internal tandem duplication (ITD)/wild type (<0.5); or CEBPA biallelic mutation]. Patients in this group will receive 2 additional courses of consolidation therapy
* Intermediate risk group [Intermediate risk cytogenetics (MRC 2010) without NPM1 mutations, FLT3-ITD, or CEBPA biallelic mutation]. Patients in this group receive an allogeneic stem cell transplant in first CR. Patients without an available donor can be autografted per center decision
* Adverse risk group [Adverse risk cytogenetics (MRC 2010), intermediate cytogenetics with FLT3-ITD without NPM1 mutation or NPM1-FLT3-ITD high ratio or MLL rearrangement; any favorable or intermediate risk patients with positive MRD following 1 (intermediate) or 2 (favorable) consolidation courses]. Intention to treat of those patients is allogeneic stem cell transplant from any source.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed AML, classified using the World Health Organization (WHO) 2017 criteria.
* Patients with 70 years old or younger.

Exclusion Criteria:

* Patients previously treated for the AML with chemotherapy different from hydroxyurea.
* Acute promyelocytic leukemia with t(15;17).
* Chronic myeloid leukemia in blastic phase.
* Secondary AML or therapy related AML.
* Presence of concomitant active neoplastic disease.
* Abnormal renal and hepatic functions with creatinin and/or bilirubin 2 times higher than the normal threshold, except when the alteration should be attributed to the leukemia.
* Patients with a cardiac ejection fraction below 45%, symptomatic cardiac deficiency or both.
* Patients with neurological or concomitant psychiatric disease.
* HIV infection.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1034 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-11-10 (Actual)

PRIMARY OUTCOMES:
Complete remission rate (CRR) | 2 months
  Analyze the efficacy and toxicity of the current doses of IC (Idarubicin and cytarabine) with G-CSF priming to achieve complete remission in patients tih AML up to 70yo.
Disease free survival (DFS) | 4 years
  Analyze the disease free survival in the whole cohort of AML patients.
Relapse rate (RR) | 4 years
  Analyze the relapse rate of all patients achieving remission with intensive induction followed by risk-adapted consolidation strategies.

SECONDARY OUTCOMES:
Feasibility of treatment completion | 4 years
  Increase the number of patients who complete all treatment phases
Survival outcome analysis of the 3 risk-adapted categories (favourable, intermediate and adverse) | 4 years
  Evaluate the feasibility of the consolidation treatments in the different risk groups by comparison of overall survival (OS), RR and DFS.
Feasibility of centralized monitoring of measurable residual disease (MRD) | 4 years
  Survival outcomes in positive vs negative MRD patients. Number of patients with modified risk due to positive MRD.
Comparison of global outcomes with previous protocol (AML-03) and other published protocols. | 4 years
  Comparison of CRR, OS, RR and DFS

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Sierra, Prof, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Jordi Esteve, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (15):
- Spain (15):
  - ICO Badalona-Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - ICO Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitari Son Espases, Palma de Mallorca, Mallorca
  - Hospital Universitari Son Llatzer, Palma de Mallorca, Mallorca
  - Hospital Verge de la Cinta, Tortosa, Tarragona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Clinic Barcelona, Barcelona
  - ICO-Girona Hopital Universitari de Girona Dr. Josep Trueta, Girona
  - Hospital Universitari Arnau de Vilanova, Lleida
  - Hospital Universitario Virgen de la Victoria, Málaga
  - ICO Tarragona-Hospital Universitari Joan XXIII, Tarragona
  - Mutua de Terrassa, Terrassa
  - Hospital Clínico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Onate G, Pratcorona M, Garrido A, Artigas-Baleri A, Bataller A, Tormo M, Arnan M, Vives S, Coll R, Salamero O, Vall-Llovera F, Sampol A, Garcia A, Cervera M, Avila SG, Bargay J, Ortin X, Nomdedeu JF, Esteve J, Sierra J; Spanish Cooperative Group for the Study and Treatment of Acute Leukemias and Myelodysplasias (CETLAM). Survival improvement of patients with FLT3 mutated acute myeloid leukemia: results from a prospective 9 years cohort. Blood Cancer J. 2023 May 5;13(1):69. doi: 10.1038/s41408-023-00839-1. PMID 37147301